CLINICAL TRIAL: NCT02310737
Title: Comparison of Postoperative Pain and Neuropathy at Cesarean Sectio With Blunt or Sharp Fascia Incision: A Prospective Randomized Controlled Double-Blinded Trial
Brief Title: Comparison of Postoperative Pain and Neuropathy at Cesarean Sectio With Blunt or Sharp Fascia Incision
Acronym: fascia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, fatma yazıcı yılmaz, medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 755
Record Dates: First submitted 2014-11-14; First posted 2014-12-08 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Postoperative Pain
Keywords: cesarean section; facial incision; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sharp incision (Active Comparator): the patients who were included as the control group (Group 1) with sharp fascia incision
  Interventions: Procedure: sharp incision
- blunt incision (Active Comparator): the patients who were included as the another group (Group 2) with blunt fascia incision
  Interventions: Procedure: blunt incision

INTERVENTIONS:
Procedure: sharp incision — The fascia will be opened with a sharp scissors in cesarean section
  Arms: sharp incision
Procedure: blunt incision — Fascia distracted from the muscle tissue with a blunt maneuver in cesarean section
  Arms: blunt incision

SUMMARY:
The purpose of this study is to compare sharp and blunt fascial entry during caesarean section.

DETAILED DESCRIPTION:
The patients will be divided into two group, The fascia will be opened with a sharp scissors in first group (group1), on the other hand in group 2 fascia distracted from the muscle tissue with a blunt maneuver. The study is planning to perform on women having cesarean section for the first time in their life and who have not previously had lower abdominal surgery before. The following parameters are evaluated for each patients

1. All patients are evaluated for postoperative pain with VAS score when they first mobilized and following postoperative1, 3 and 7 days; 1 and 3 months 2. Postoperative sensory loss on skin incision scar, lower abdomen, pelvic region, groin, inner thigh, and labia majus

ELIGIBILITY:
Inclusion Criteria:

* Woman having caesarean section for the first time
* Woman, who have had no previous lower abdominal surgery
* Woman who can give informed consent

Exclusion Criteria:

Diabetes Mellitus (This does not include gestational diabetes)

* Infection
* Regular treatment with immunosuppressives
* Alcohol or drug abuse
* Age under 18 years old
* Chronic pain disease eg. fibromyalgia, rheumatoid arthritis
* BMI over 35

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
postoperative pain scores change on the Visual Analog Scale (VAS) | 1, 3 and 7 days
  the difference in pain scores between two groups 1, 3 and 7 days postoperatively. Pain is registered by a score on a vas-scale from 0-10.Changes on VAS scale reported.

SECONDARY OUTCOMES:
postoperative sensory loss change on skin incision scar, lower abdomen, pelvic region, groin, inner thigh, and labia majus | 7 days postoperatively
  assessment of the sensory loss difference on skin incision scar, lower abdomen, pelvic region, groin, inner thigh, and labia majus postoperatively(day7). Sensory loss measured by asking their sensory feelings on scar area, lower abdomen, pelvic region, groin, inner thigh, and labia majus
postoperative pain scores change on the Visual Analog Scale (VAS) | 1and 3 months postoperatively
  the difference in pain scores between two groups 1 and 3 months postoperatively. Pain is registered by a score on a vas-scale from 0-10.
postoperative sensory loss change on skin incision scar | 1and 3 months postoperatively
  Assessment of the sensory loss difference on skin incision scar, lower abdomen, pelvic region, groin, inner thigh, and labia majus postoperatively at 1 and 3 months. Sensory loss measured by asking their sensory feelings on scar area, lower abdomen, pelvic region, groin, inner thigh, and labia majus

CONTACTS AND LOCATIONS:
Overall Officials: fatma yazıcı yılmaz, md, Principal Investigator — sisli etfal training research and hospital
Locations (1):
- Fatma Yazıcı Yılmaz, Istanbul, Turkey (Türkiye)